CLINICAL TRIAL: NCT04349410
Title: The Fleming [FMTVDM] Directed CoVid-19 Treatment Protocol
Acronym: FMTVDM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Camelot Foundation (Other)
Responsible Party: Principal Investigator, RM Fleming, MD, Principle Investigator, The Camelot Foundation
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: FMTVDM2020
Record Dates: First submitted 2020-04-11; First posted 2020-04-16 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: CoVid 19 Positive
MeSH Terms: interventions — Hydroxychloroquine; Azithromycin; Doxycycline; Clindamycin; Primaquine; remdesivir; tocilizumab; Methylprednisolone; Interferon-alpha2b; Losartan; COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Measurement of CoVid-19 pneumonia (CVP) and inflammation will be made using a patented method (FMTVDM #9566037 and adjunct USPTO submissions deemed covered by USPTO under the original patent #9566037).
  Following FMTVDM measurements, patients will be randomized into one of eleven treatment arms - others may be added as information becomes available. Forty-eight to 72-hours later - providing adequate time for treatment effect - FMTVDM will be repeated.
  Patients with improvement in FMTVDM will be maintained on their original treatment. FMTVDM measured treatment failure will result in a change to another arm of treatment. FMTVDM measurement showing no change will be treated by adding an additional treatment arm to patient care. Sequential FMTVDM studies will be carried out.
  Simultaneous Immune and ventilatory RX. Ventilatory support per ARDS protocol. Applicable blood tests and PCR will be included.
Who Masked: Investigator
Masking Description: As FMTVDM is an absolute quantification method, which cannot be influenced by human error or bias, the final determinant of success or failure of treatment cannot be influenced. However, given the pandemic, medical, nursing, technologist and other healthcare providers will NOT be blinded to data. The availability of the data will allow real time assessment and decision making by the clinicians involved in the care of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- Treatment 1 (Experimental): Hydroxychloroquine 200 mg po q 8 hrs (600 mg qD) for a total of 10-days OR Hydroxychloroquine 155 mg IV every 8-hours (600 mg qD) for 10-days if patient is intubated and Azithromycin 500 mg IV on day 1, followed by 250 mg IV on days 2-5 (to prevent bacterial superinfection ).
  Interventions: Drug: Hydroxychloroquine, Azithromycin
- Treatment 2 (Experimental): Hydroxychloroquine 200 mg po q 8 hrs (600 mg qD) for a total of 10-days OR Hydroxychloroquine 155 mg IV every 8-hours (600 mg qD) for 10-days if patient is intubated and Doxycycline 100mg IV q 12 hrs with each dose given over 1 to 4-hours (to prevent bacterial superinfection ).
  Interventions: Drug: Hydroxychloroquine, Doxycycline
- Treatment 3 (Experimental): Hydroxychloroquine 200 mg po q 8 hrs (600 mg qD) for a total of 10-days OR Hydroxychloroquine 155 mg IV every 8-hours (600 mg qD) for 10-days if patient is intubated Clindamycin 150-450 mg po q6 hours x 10 days OR 4800 mg IV daily - beginning with 150 mg initial rapid infusion, followed by continuous infusion q 24-hours for 7-days.
  Interventions: Drug: Hydroxychloroquine, Clindamycin
- Treatment 4 (Experimental): Hydroxychloroquine 200 mg po q 8 hrs (600 mg qD) for a total of 10-days OR Hydroxychloroquine 155 mg IV every 8-hours (600 mg qD) for 10-days if patient is intubated Primaquine 200 mg po on day # 1. Clindamycin 150-450 mg po q6 hours x 10 days OR 4800 mg IV daily - beginning with 150 mg initial rapid infusion, followed by continuous infusion q 24-hours for 7-days.
  Interventions: Drug: Hydroxychloroquine, Clindamycin, Primaquine - low dose.
- Treatment 5 (Experimental): Primaquine 200 mg po on day # 1. Clindamycin 150-450 mg po q6 hours x 10 days OR 4800 mg IV daily - beginning with 150 mg initial rapid infusion, followed by continuous infusion q 24-hours for 7-days. This treatment arm is not available for intubated patients due to the absence of an IV form of Primaquine.
  Interventions: Drug: Hydroxychloroquine, Clindamycin, Primaquine - high dose.
- Treatment 6 (Experimental): Remdesivir 200 mg IV on day 1, followed by 100 mg IV qD for a total of 10-days.
  Interventions: Drug: Remdesivir
- Treatment 7 (Experimental): Tocilizumab 8mg/kg IV (not to exceed 800 mg) over 60-minutes. If clinical improvement is not noted, three additional doses may be administered at q 8-hour intervals from the initial infusion for a total of 4-doses maximum.
  ANY PATIENT DEMONSTRATING CYTOKINE RELEASE SYNDROME WILL HAVE THIS TREATMENT ARM AUTOMATICALLY ADDED.
  Interventions: Drug: Tocilizumab
- Treatment 8 (Experimental): Methylprednisolone 125 mg IV every 6-hours for 3 days; then 125 mg IV every 12-hours for 2 days; then 125 mg IV daily for 2 days; then 60 mg IV daily for 2 days [with each infusion given over 30-minutes]; then Solumedrol dose pack to taper off steroids.
  Interventions: Drug: Methylprednisolone
- Treatment 9 (Experimental): Interferon alpha-2b 5 million units per nebulizer BID.
  Interventions: Drug: Interferon-Alpha2B
- Treatment 10 (Experimental): Losartan 25 mg po qD. IRB held due to questions about benefit.
  Interventions: Drug: Losartan
- Treatment 11 (Experimental): Convalescent Plasma 2-units ABO-compatible with antibody titer of 1:320 dilution. Each unit intravenously infused over 4-hours.
  Interventions: Drug: Convalescent Serum

INTERVENTIONS:
Drug: Hydroxychloroquine, Azithromycin — FMTVDM Planar, SPECT, PET
  Arms: Treatment 1
Drug: Hydroxychloroquine, Doxycycline — FMTVDM Planar, SPECT, PET
  Arms: Treatment 2
Drug: Hydroxychloroquine, Clindamycin — FMTVDM Planar, SPECT, PET
  Arms: Treatment 3
Drug: Hydroxychloroquine, Clindamycin, Primaquine - low dose. — FMTVDM Planar, SPECT, PET
  Arms: Treatment 4
Drug: Hydroxychloroquine, Clindamycin, Primaquine - high dose. — FMTVDM Planar, SPECT, PET
  Arms: Treatment 5
Drug: Remdesivir — FMTVDM Planar, SPECT, PET
  Arms: Treatment 6
Drug: Tocilizumab — FMTVDM Planar, SPECT, PET
  Arms: Treatment 7
Drug: Methylprednisolone — FMTVDM Planar, SPECT, PET
  Arms: Treatment 8
Drug: Interferon-Alpha2B — FMTVDM Planar, SPECT, PET
  Arms: Treatment 9
Drug: Losartan — FMTVDM Planar, SPECT, PET
  Arms: Treatment 10
Drug: Convalescent Serum — FMTVDM Planar, SPECT, PET
  Arms: Treatment 11

SUMMARY:
Diagnostic determination of disease and treatment responses has been limited to qualitative imaging, measurement of serum markers of disease, and sampling of tissue. In each of these instances, there is a built in error either due to sensitivity and specificity issues, clinician interpretation of results, or acceptance of the use of an indirect marker (blood test) of what is happening elsewhere in the body - at the tissue level.

The Fleming Method for Tissue and Vascular Differentiation and Metabolism (FMTVDM) using same state single or sequential quantification comparisons [1] provides the first and only patented test (#9566037) - along with the associated submitted patent applications ruled to be covered under #9566037 - that quantitatively measures changes in tissue resulting from inter alia a disease process. This includes inter alia coronary artery disease (CAD), cancer and infectious/inflammatory processes including CoVid-19 pneumonia (CVP) resulting from the metabolic and regional blood flow differences (RBFDs) caused by these diseases.

The purpose of this paper is to make clinicians and researchers aware of this proposed method for investigating the prevalence and severity of CVP - in addition to providing rapid determination of treatment response in each patient, directing treatment decisions; thereby reducing the loss of time, money, resources and patient lives.

DETAILED DESCRIPTION:
FMTVDM - See Appendix A.

1. Quantitatively calibrates the nuclear camera to guarantee that the measurements made by the camera are accurate, consistent and reproducible. This quantification is dependent upon the isotope being used, the camera and the timing sequence of image acquisition. Such calibration is NOT currently done and it is part of the patent. Studies have demonstrated that the lack of this quantitative calibration has resulted in up to 1/3 of the data being lost for SUV and qualitative interpretation; in addition to making quantification impossible.
2. The patient presents in a fasting state - to eliminate digestive processes from interfering with blood flow distributions - and the differences in metabolic and regional blood flow differences (RBFDs) are enhanced with vasodilatory agents, shifting blood flow and isotope towards regions of greater blood flow and metabolism; enhancing isotope delivery, uptake and quantification.
3. With a now quantitatively calibrated nuclear camera - in this instance a PLANAR camera - or SPECT/CT or PET/CT/MRI if specifically approved - to allow imaging to be done at patient's bedside reducing the use of hospital resources required for transport and decrease potential for patient complications resulting from a transport - image acquisition will occur for 10-minutes following peak enhancement effect of the vasodilatory agent and timed injection of the isotope based upon the enhancing agent.

   Regions-of-interest (ROIs) will drawn by the nuclear technologist - either at the bedside or in the nuclear laboratory - to provide FMTVDM measurements using software already present in the nuclear camera systems. Specific ROIs will be drawn of the right lung (total), left lung (total), mediastinum (thymus activity), and any specific areas where increased tracer uptake is noted.
4. These FMTVDM measurements including MAXIMAL COUNTS +/- VARIANCE, provide the values of the most active pulmonary tissue resulting from the CoVid-19 infection and inflammatory response; just as it has previously been used for CAD and Cancer.
5. From these FMTVDM measurements, the pulmonary tissue and the CoVid-19 infectious process results are placed on a Health-Spectrum showing where in the tissue transitioning process the patient is. The measurements also provide information about how rapidly the tissue is changing. FMTVDM provides the quantitative measurement of where the patient is at any point in time during their course of treatment and how they compare with other patients.
6. Once the FMTVDM measurements have been obtained, treatment decisions can be made based upon serial changes in FMTVDM. Treatments outcomes are based upon FMTVDM measurements, including the maximum FMTVDM and the variance in those measurements. By comparing serial FMTVDM results, improvement or deterioration in the patient's health and the success or failure of the current treatment regimen is measured, providing patient-centered, patient-specific, patient-oriented and patient-directed decisions. Thus saving time, money, resources and lives - not to mention unnecessary side effects from treatment, which is not working.

ELIGIBILITY:
Inclusion Criteria: CoVid-19 -

Exclusion Criteria: Decision by patient to not participate.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2020-04-11 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Improvement in FMTVDM Measurement with nuclear imaging. | 72 hours
  Measured improvement in tissue as measured using FMTVDM

SECONDARY OUTCOMES:
Ventilator status | 7 days
  Extubation
Survival status | 30 days
  Self explanatory

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Fleming, PhD, MD, JD, Study Chair — FHHI-OI-Camelot;QME
Locations (1):
- FHHI-OI-Camelot; QME, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through electronic request from approved individuals and institutions.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This will depend upon the availability of staff given the multi-nation approach to this project.
Access Criteria: Expressed request through email as listed.

REFERENCES:
- See also: FMTVDM Patent # 9566037 — https://patents.google.com/patent/US9566037B2/en
- See also: The Critical Importance of Quantifying Tissue Change instead of using qualitative or semi-quanitified results. — https://rdcu.be/b22Dd
- See also: FMTVDM quantification for coronary artery disease and inflammation — https://www.novapublishers.com/catalog/product_info.php?products_id=8409
- See also: FMTVDM quantification. — https://www.mdedge.com/fedprac/issue/73998/federal-practitioner-276
- See also: Infection and Inflammation reversal by treatment of pathogens with associated reductions in IL-6. — https://www.ncbi.nlm.nih.gov/pubmed/10667648

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04349410/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04349410/ICF_002.pdf